CLINICAL TRIAL: NCT03881371
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Safinamide, as add-on Therapy, in Idiopathic Chinese Parkinson's Disease (PD) Patients With Motor Fluctuations Treated With Stable Doses of Levodopa
Brief Title: A Study to Evaluate the Efficacy and Safety of Safinamide, as add-on Therapy, in Idiopathic Chinese Parkinson's Disease (PD) Patients With Motor Fluctuations Treated With Stable Doses of Levodopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z7219L05
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safinamide (Experimental): Patient will receive film-coated Safinamide tablets orally at an initial dose of 50 mg once daily (OD) and then will be increased the day after the Visit 3/week 2 (ideally at day 15) to the final dose of 100 mg OD. Treatment will continue daily for a total of 16 weeks.
  Interventions: Drug: Safinamide
- Placebo (Placebo Comparator): Patient will receive matching placebo orally at an initial dose of 50 mg once daily (OD) and then will be increased the day after the Visit 3/week 2 (ideally at day 15) to the final dose of 100 mg OD. Treatment will continue daily for a total of 16 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Safinamide — At baseline (Day 1), eligible patients will be randomised to receive safinamide (initial 50 mg titrated to 100 mg the day after the Visit 3/week 2, ideally at day 15). The investigational medicinal product (IMP) will be taken in the morning at breakfast time, in addition to the morning dose of L-dopa and other (if any) PD medications.
  Arms: Safinamide
Other: Placebo — At baseline (Day 1), eligible patients will be randomised to receive matching placebo, orally OD. Placebo will be added to the standard stabilized treatment as a control of the safinamide group, hence patients on placebo will have benefit from other ongoing anti-PD medication
  Arms: Placebo

SUMMARY:
This is a Phase III, multicentre, randomised, double-blind, placebo-controlled study to evaluate the effects of 100 mg safinamide, administered orally once daily (OD), in Chinese Parkinson's disease (PD) patients, experiencing motor fluctuations while on stable doses of Levodopa (L-dopa) (alone or in combination with other anti-Parkinson drugs). Eligible patients are required to meet the United Kingdom PD Society Brain Bank Clinical Diagnostic Criteria. The study involves a placebo group. Placebo will be added to the standard stabilized treatment as a control of the safinamide group, hence patients on placebo will have benefit from other ongoing anti-PD medication. A total of 306 patients will be randomised into this study (153 in the safinamide and 153 in the placebo groups).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years old.
2. Chinese ethnicity.
3. Able to understand and willing to provide written informed consent.
4. Able to maintain an accurate and complete 24-hour diary with the help of a caregiver.
5. Diagnosis of idiopathic Parkinson's Disease (IPD) using the United Kingdom Parkinson's Disease Society Brain Bank criteria of more than 3 years duration.
6. Be levodopa responsive and receiving treatment with stable daily doses of oral L-dopa, with or without benserazide/carbidopa, with or without addition of a catechol-O-methyltransferase (COMT) inhibitor and may be receiving concomitant treatment with stable doses of dopamine agonists, anticholinergics and/or amantadine for at least 4 weeks prior to the screening visit.
7. A Hoehn and Yahr stage between 1-4 inclusive during the "ON" phase.
8. Experiencing motor fluctuations with a minimum of 1.5 hours/day of "OFF" time during the day (excluding morning akinesia), based on historical data.
9. If female, be post-menopausal for at least one year or have undergone hysterectomy or, if of child-bearing potential, must have a negative pregnancy test, must not be breast-feeding nor become pregnant during the study and must use adequate contraception for 1 month prior to randomisation and for up to 1 month after the last dose of study drug. Adequate contraception is defined as:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives or a non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit;
   2. a male sexual partner who agrees to use a male condom with spermicide or a sterile sexual partner . For all women of child-bearing potential, urine pregnancy test result at screening must be negative.

For all women of child-bearing potential, urine pregnancy test result at screening must be negative.

Exclusion Criteria:

1. Any form of Parkinsonism other than IPD.
2. Diagnosis of chronic migraine (>15 days per month) or cancer pain.
3. L-dopa infusion.
4. Hoehn and Yahr stage 5 during the "ON" phase.
5. If female, pregnancy or breast-feeding.
6. Neurosurgical intervention of PD or stereotactic brain surgery.
7. Severe peak dose or biphasic dyskinesia, unpredictable or widely swinging fluctuations.
8. History of major depression or other clinically significant psychotic disorder which compromise the ability to provide the informed consent or to participate to the study.
9. Drug and/or alcohol abuse within 12 months prior to the screening visit.
10. History of dementia or severe cognitive dysfunction.
11. Use of any investigational drug or device within 30 days prior to screening or 5 half-lives, whichever is the longest, or during the study.
12. Allergy/sensitivity or contraindications to the investigational medicinal products (IMPs) or their excipients, to anticonvulsants or to anti-Parkinson drugs.
13. Any clinically significant condition (including laboratory values) which, in the opinion of the Investigator, would not be compatible with study participation or represent a risk for patients while in the study.
14. Moderate or severe liver failure using the Child-Pugh classification score, or human immunodeficiency virus (HIV) infection.
15. Treatment with monoamine oxidase inhibitors (MAOIs), pethidine, opiates, opioids, fluoxetine, fluvoxamine in the 4 weeks prior to the screening visit. These drugs are not allowed throughout the study and up 2 weeks after the last dose of study drug.
16. Ophthalmologic history including any of the following conditions: albinism, uveitis, retinitis pigmentosa, retinal degeneration, active retinopathy, severe progressive diabetic retinopathy, inherited retinopathy or family history of hereditary retinal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Sir Run Run Shaw Hospital, Zhejiang University 浙江大学医学院附属邵逸夫医院, Hangzhou, No 3, Qing Chun East Road
  - Shanghai Ninth People's Hospital 上海交通大学医学院附属第九人民医院, Shanghai, No 639, Zhizaoju Road
  - Tianjin Union Medicine Center 天津市人民医院, Tianjin, No. 130, Jie Yuan Rd., Hong Qiao District
  - The Third Xiangya Hospital of Central South University 中南大学湘雅三医院, Changsha, No. 138, Tong Zi Po Road, He XI Yue Lu District
  - Renmin Hospital of Wuhan University 武汉大学人民医院, Wuhan, No. 238, Jie Fang Road
  - Sichuan Provincial People's Hospital 四川省医学科学院·四川省人民医院, Chengdu, No. 32 XI Er Duan, First Ring Road, Qing Yang District
  - West China Hospital, Sichuan University 四川大学华西医院, Chengdu, No. 37, Guoxue Alley
  - Beijing Friendship Hospital 首都医科大学附属北京友谊医院, Beijing, No. 6, Tiantan XI Li, Chongwen District
  - Beijing Tiantan Hospital Affiliated to Capital Medical University 首都医科大学附属北京天坛医院, Beijing, No. 6, Tiantan XI Li, Chongwen District
  - The First Bethune Hospital of Jilin University, Changchun, No. 71, Xin Min Street
  - The First Hospital of Shanxi Medical University 山西医科大学第一医院, Taiyuan, No. 85, Jie Fang South Road
  - The Second Affiliated Hospital of Zhejiang University 浙江大学医学院附属第二医院, Hangzhou, No. 88, Jie Fang Rd.
  - The Second Affiliated Hospital of Nanchang University 南昌大学第二附属医院, Nanchang, No.1 Minde Road of Nanchang
  - Guangzhou First People's Hospital 广州市第一人民医院, Guangzhou, No.1 Panfu Rd.
  - Shanghai General Hospital 上海市第一人民医院, Shanghai, No.100 Haining Road
  - Sun Yat-sen Memorial Hospital 中山大学孙逸仙纪念医院, Guangzhou, No.107, Yanjiang West Road
  - Tongji Hospital of Tongji University 同济大学附属同济医院, Wuhan, No.1095 Jiefang Avenue
  - The Third Hospital of Hebei Medical University 河北医科大学第三医院, Shijiazhuang, No.139.Zi Qiang Rd
  - Chongqing Three Gorges Central Hospital 重庆三峡中心医院, Chongqing, No.165 Xincheng Rd, Wanzhou District
  - Shanghai Ruijin Hospital 上海交通大学医学院附属瑞金医院, Shanghai, No.197 Ruijin Er Road
  - The First Affiliated Hospital of Baotou Medical University 内蒙古科技大学包头医学院第一附属医院, Baotou, No.41 Linyin Road
  - Baotou City Central Hospital 包头市中心医院, Baotou, No.61, Huancheng Road, Donghe District
  - The Affiliated Hospital of Xuzhou Medical University 徐州医科大学附属医院, Xuzhou, No.99, Huaihai West Road, Xuzhou, Jiangsu
  - The Affiliated Hospital Of Guiyang Medical College 贵州医科大学附属医院, Guiyang, No28. Guiyi Street
  - The First Affiliated Hospital of Guangzhou Medical University 广州医科大学附属第一医院, Guangzhou, Number 151, Yanjiang Road
  - Wenzhou Medical College-The First Affiliated Hospital 温州医科大学附属第一医院, Wenzhou, Shangcai Burg, Ouhai District
  - Daqing Oilfield General Hospital 大庆油田总医院, Daqing
  - Fujian Medical University Union Hospital 福建医科大学附属协和医院, Fuzhou
  - Qilu Hospital of Shandong University 山东大学齐鲁医院, Jinan
  - Nanjing Drum Tower Hospital 南京鼓楼医院, Nanjing
  - The second affiliated hospital of Soochow University 苏州大学附属第二医院, Suzhou

REFERENCES:
- [Derived] Dei Cas A, Micheli MM, Aldigeri R, Gardini S, Ferrari-Pellegrini F, Perini M, Messa G, Antonini M, Spigoni V, Cinquegrani G, Vazzana A, Moretti V, Caffarra P, Bonadonna RC. Long-acting exenatide does not prevent cognitive decline in mild cognitive impairment: a proof-of-concept clinical trial. J Endocrinol Invest. 2024 Sep;47(9):2339-2349. doi: 10.1007/s40618-024-02320-7. Epub 2024 Apr 2. PMID 38565814
- [Derived] Cattaneo C, Kulisevsky J. The Effects of Safinamide in Chinese and Non-Chinese Patients with Parkinson's Disease. Adv Ther. 2024 Feb;41(2):638-648. doi: 10.1007/s12325-023-02736-2. Epub 2023 Dec 9. PMID 38070039
- [Derived] Wei Q, Tan Y, Xu P, Tao E, Lu Z, Pan X, Wang B, Liu C, Dong X, Tian Y, Sun X, Cattaneo C, Chen S, Shang H; XINDI Study Investigators Group. The XINDI Study: A Randomized Phase III Clinical Trial Evaluating the Efficacy and Safety of Safinamide as Add-On Therapy to Levodopa in Chinese Patients with Parkinson's Disease with Motor Fluctuations. CNS Drugs. 2022 Nov;36(11):1217-1227. doi: 10.1007/s40263-022-00958-6. Epub 2022 Nov 8. PMID 36346534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 307 patients were randomized at approximately 31 study centres in China between 01-Aug-2019 to 20-Aug-2021.
Pre-assignment Details: Patients who met the inclusion and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment. The study was composed of a screening period (up to 2 weeks prior to the start of treatment, with 1 screening visit) and a treatment period (16 weeks).
Groups:
- Safinamide: Patients received film-coated Safinamide tablets orally, once daily (od) with L-dopa and other (if any) anti-Parkinson drugs. After the Week 2 (ideally at Day 15), the dosage was adjusted from 50 mg to 100 mg and was maintained at 100 mg until the end of the study. Treatment continued daily for a total of 16 weeks.
- Placebo: Patients received matching placebo orally, od with L-dopa and other (if any) anti-Parkinson drugs. After the Week 2 (ideally at Day 15), the dosage was adjusted from 50 mg to 100 mg and was maintained at 100 mg until the end of the study. Treatment continued daily for a total of 16 weeks.
Period: Overall Study
Arm/Group | Safinamide | Placebo
Started | 153 (2 patients randomized in error due to failure to meet inclusion criteria, and were not treated. 1 patient complete early termination visit with end of treatment (EOT) status, and other prematurely withdraw from the study immediately without EOT status.) | 154
Number Treated | 151 | 154
Completed | 137 | 130
Not Completed | 16 | 24
Not completed — Adverse Event | 8 | 9
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-Compliance with Study Drug | 0 | 2
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 2 | 10
Not completed — Discontinuation from Study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population were included all patients who provided informed consent and received at least 1 dose or partial dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safinamide | Placebo | Total
Number analyzed (Participants) | 151 | 154 | 305
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (9.29) | 61.8 (9.28) | 61.6 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 69 | 128
  Male | 92 | 85 | 177
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 151 | 154 | 305

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in the Mean Total Daily "OFF" Time
Description: The mean total daily "OFF" time was assessed by 24-hour patient diary cards, of safinamide 100 mg/day compared to placebo, given as add-on therapy in PD patients with motor fluctuations on stable doses of L-dopa. Patients completed the daily diary by selecting one of the following five options for each 30-minute time period:
  * "OFF" (Stiffness, marked decrease in mobility, or immobility).
  * "ON" without dyskinesia (Good or practically normal mobility without dyskinesia).
  * "ON" with non-troublesome dyskinesia (With dyskinesia but it does not interfere with function/cause meaningful discomfort).
  * "ON" with troublesome dyskinesia (With dyskinesia which interferes with function/causes meaningful discomfort. Of note, these dyskinesia movements are different from the rhythmic "tremor" (a symptom of Parkinson's Disease itself).
  * Asleep (Time spent asleep).
Time Frame: At baseline and Week 16
Population: Full analysis set population (FAS) included all patients who provided informed consent, were randomized and received at least 1 dose or partial dose of the study drug.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 151 | 154
Hours | -1.93 (2.556) | -0.88 (2.543)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p < .0001, ANCOVA — Analysis was based on a covariance model (ANCOVA) with treatment and centre as independent factors, baseline mean total daily "OFF" time measurement as covariate and change from baseline as dependent variable; Least-Square Mean = -1.10, 95% CI 2-sided [-1.643 to -0.555], Standard Error of Mean 0.277

2. Secondary Outcome: Change From Baseline to Week 16 in Pain Severity, as Assessed by an 11 Point Numerical Rating Scale (NRS)
Description: The pain severity, was assessed by an 11-point Numerical Rating Scale (NRS). The NRS is a segmented numeric version of the visual analogue scale (VAS) in which a patient selects a whole number that best reflects the intensity of his/her pain, ranging from '0' ("no pain") to '10' ("worst possible pain").
Time Frame: At baseline and Week 16
Population: The FAS population included all patients who provided informed consent, were randomized and received at least 1 dose or partial dose of the study drug.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 151 | 154
Score on a Scale | -0.0 (1.89) | -0.0 (2.14)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p = 0.8901, ANCOVA — ANCOVA with treatment and centre as independent factors, baseline NRS measurement as covariate and change from baseline as dependent variable; Least-Square Mean = -0.03, 95% CI 2-sided [-0.440 to 0.382], Standard Error of Mean 0.210

3. Secondary Outcome: Change From Baseline to Week 16 in the Mean Total Daily "ON" Time
Description: The mean total daily "ON" time, as assessed by 24-hour patient diary cards. Patients completed the daily diary by selecting one of the following five options for each 30-minute time period:
  * "OFF" (Stiffness, marked decrease in mobility, or immobility).
  * "ON" without dyskinesia (Good or practically normal mobility without dyskinesia).
  * "ON" with non-troublesome dyskinesia (With dyskinesia but it does not interfere with function/cause meaningful discomfort).
  * "ON" with troublesome dyskinesia (With dyskinesia which interferes with function/causes meaningful discomfort. Of note, these dyskinesia movements are different from the rhythmic "tremor" (a symptom of Parkinson's Disease itself).
  * Asleep (Time spent asleep).
Time Frame: At baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 137 | 130
Hours | 1.30 (2.693) | 0.51 (2.875)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p = 0.0049, ANCOVA — ANCOVA with treatment and centre as independent factors, baseline mean total daily "ON" time measurement as covariate and change from baseline as dependent variable; Least-Square Mean = 0.89, 95% CI 2-sided [0.274 to 1.515], Standard Error of Mean 0.315

4. Secondary Outcome: Change From Baseline to Week 16 in the Mean Daily "ON" Time With no/Non Troublesome Dyskinesia
Description: The mean daily "ON" time with no/non troublesome dyskinesia, as assessed by 24-hour patient diary cards. Patients completed the daily diary by selecting one of the following five options for each 30-minute time period:
  * "OFF" (Stiffness, marked decrease in mobility, or immobility).
  * "ON" without dyskinesia (Good or practically normal mobility without dyskinesia).
  * "ON" with non-troublesome dyskinesia (With dyskinesia but it does not interfere with function/cause meaningful discomfort).
  * "ON" with troublesome dyskinesia (With dyskinesia which interferes with function/causes meaningful discomfort. Of note, these dyskinesia movements are different from the rhythmic "tremor" (a symptom of Parkinson's Disease itself).
  * Asleep (Time spent asleep).
Time Frame: At baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 137 | 130
Hours | 1.30 (2.927) | 0.39 (3.212)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Test type: Superiority; p = 0.0021, ANCOVA — ANCOVA with treatment and centre as independent factors, baseline mean total daily "ON" time with no/non-troublesome Dyskinesia measurement as covariate and change from baseline as dependent variable; Least-Square Mean = 1.07, 95% CI 2-sided [0.392 to 1.753], Standard Error of Mean 0.345

5. Secondary Outcome: Change From Baseline to Week 16 in the Unified Parkinson's Disease Rating Scale (UPDRS) Total Score During the "ON" Phase
Description: The UPDRS comprises 3 parts that evaluates any complication of treatment: Part I: Evaluation of mentation or cognition, behavior and mood. Part II: Evaluation of the activities of daily life. Part III: Evaluation of motor function. Part IV: Evaluation of complications of therapy. The UPDRS performed by the Investigator with points assigned to each item in the scale based on the patient's response as well as observation and physical examination. Together Parts I-III contain 44 items, with each item scored on a 5-point scale. Part IV contains 11 questions with a scale ranging from 0 to 23. Thus, the final total score may range from 0 (no disability) to 199 (total disability). The UPDRS is the most commonly used scale in clinical studies to follow the longitudinal course of PD. Part I Evaluation of mentation or cognition, behavior and mood contains 4 items with each item scored on a 5 point scale, the scale ranging from 0 to 16.
Time Frame: At baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 134 | 128
Change in score | -12.3 (13.59) | -5.8 (12.30)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p < .0001, ANCOVA — ANCOVA with treatment and centre as independent factors, baseline UPDRS score as covariate and change from baseline as dependent variable; Least-Square Mean = -5.99, 95% CI 2-sided [-8.842 to -3.141], Standard Error of Mean 1.447

6. Secondary Outcome: Change From Baseline to Week 16 in the UPDRS Part II Activities of Daily Living (ADL) Score During the "ON" Phase
Description: The UPDRS= Unified Parkinson's Disease Rating Scale; is the most commonly used scale in clinical studies to follow the longitudinal course of PD.
  It is divided in 4 sections, each of them with several items. The score of each item is 0-1 or 0-4 (the majority) where 0 is no symptom while the highest score means the most severe symptom.
  UPDRS part I: 4 items, score 0-16 (total); UPDRS part II: 13 items, score 0-52 (total); UPDRS part III: 14 items, score 0-108 (total) UPDRS part IV: it is dived in 3 sections. Section A=dyskinesias, 4 items, score 0-13 (total); section B=clinical fluctuations, 4 items, score 0-7 (total); section C=other complications, 3 items, score 0-3 (total).
  The total score of the UPDRS (meaning of all the 4 parts) is 0-199 where 0 means no symptoms, 199 the most severe symptoms.
Time Frame: At baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 134 | 128
Change in score | -2.7 (4.45) | -1.2 (4.32)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p = 0.0033, ANCOVA — ANCOVA with treatment and centre as independent factors, baseline UPDRS part II (ADL) score as covariate and change from baseline as dependent variable; Least-Square Mean = -1.52, 95% CI 2-sided [-2.521 to -0.511], Standard Error of Mean 0.510

7. Secondary Outcome: Change From Baseline to Week 16 in the UPDRS Part III (Motor Function) Score During the "ON" Phase
Description: as for outcome 6
Time Frame: At baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 134 | 128
Change in score | -8.2 (9.64) | -3.7 (8.71)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p = 0.0002, ANCOVA — ANCOVA with treatment and centre as independent factors, baseline UPDRS part III (motor function) score as covariate and change from baseline as dependent variable; Least-Square Mean = -3.80, 95% CI 2-sided [-5.749 to -1.856], Standard Error of Mean 0.988

8. Secondary Outcome: Clinical Global Impression of Severity (CGI-S) Score Assessed at Week 16
Description: The CGI-S scale measures global severity of illness at a given point in time. It is rated on a 7-point Likert-type scale ranging from 1 (normal, not ill at all) to 7 (extremely severe). The CGI-S was assessed at all visits, starting at baseline.
Time Frame: At week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Point on scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 134 | 128
Point on scale | 3.6 (0.80) | 3.8 (0.95)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p = 0.0150, Wilcoxon (Mann-Whitney) — Analysis was based on the Wilcoxon-Mann-Whitney test stratified by centre; Median = 0.0, 95% CI 2-sided [0.000 to 0.000] — Non-parametric 95% confidence interval was presented for the treatment difference in CGI-S at each post-baseline visit as reported by the Hodges-Lehmann estimator

9. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Assessed at Week 16
Description: The CGI-C scale measured the change in the patient's clinical status from baseline using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change. The change from the patient's baseline condition is assessed by the Investigator at all post-baseline visits.
Time Frame: At baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Point on scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 134 | 128
Point on scale | 3.0 (1.12) | 3.4 (1.03)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p = 0.0007, Wilcoxon (Mann-Whitney) — Analysis was based on the Wilcoxon-Mann-Whitney test stratified by centre; Median = 0.5, 95% CI 2-sided [0.000 to 1.000] — Non-parametric 95% confidence interval was presented for the treatment difference in CGI-C score at each post-baseline visit as reported by the Hodges-Lehmann estimator

10. Secondary Outcome: Change From Baseline to Week 16 in the Parkinson's Disease Questionnaire-39 Items (PDQ-39) Score
Description: The PDQ-39 comprises 39 questions measuring eight dimensions of health: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily pain. Dimension scores are coded on a scale of 0 (perfect health as assessed by the measure) to 100 (worst health as assessed by the measure).
Time Frame: At baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 134 | 128
Change in score | -6.42 (10.223) | -2.67 (10.901)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; Treatment difference (Safinamide - Placebo); Test type: Superiority; p = 0.0033, ANCOVA — ANCOVA with treatment and centre as independent factor, baseline Summary Index score as covariate and change from baseline as dependent variable; Least-Square Mean = -3.36, 95% CI 2-sided [-5.589 to -1.128], Standard Error of Mean 1.132

11. Other Pre Specified Outcome: Number of Patients With Treatment-emergent Adverse Events (TEAE) and Treatment-emergent Serious Adverse Event (TESAE)
Description: Evaluation of the safety and tolerability of safinamide compared with placebo in Chinese PD patients with motor fluctuations.
Time Frame: From baseline until follow-up visit (1 Week after the end of treatment [Up to 2 Years])
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 151 | 154
Participants
  Any TEAE | 105 | 88
  Any TEAE Related to study drug | 54 | 40
  Any Severe TEAE | 4 | 4
  Any Severe TEAE, Related to study drug | 3 | 1
  Any TEAE with Outcome of Death | 1 | 0
  Any TEAE with Outcome of Death to study drug | 1 | 0
  Any TESAE | 8 | 5
  Any TESAE, Related to Study Drug | 4 | 3
  Any TEAE Leading to Study Withdrawal | 8 | 9
  Any TEAE Leading to Discontinuation of Study Drug | 8 | 10
  Any TESAE Leading to Study Withdrawal | 3 | 1
  Any TESAE Leading to Discontinuation of Study Drug | 3 | 1
  Any TEAE Leading to Discontinuation of Study Drug | 7 | 10
  Any TEAE Leading to Dose Reduction of Study Drug | 7 | 2

ADVERSE EVENTS:
Time Frame: From baseline until follow-up visit (1 Week after the end of treatment [Up to 2 Years])
Arm/Group | Safinamide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/151 | 0/154
Serious Adverse Events (participants affected / at risk) | 8/151 | 5/154
Other Adverse Events (participants affected / at risk) | 42/151 | 35/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safinamide (N=151) | Placebo (N=154)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Vascular headache (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safinamide (N=151) | Placebo (N=154)
Dyskinesia (Nervous system disorders) | 18 (18) | 6 (6)
Dizziness (Nervous system disorders) | 9 (15) | 10 (14)
Parkinson's disease (Nervous system disorders) | 7 (7) | 14 (15)
Constipation (Gastrointestinal disorders) | 6 (6) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03881371/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03881371/SAP_001.pdf